CLINICAL TRIAL: NCT01694186
Title: A Phase III, Multi-National, Multi-Center, Randomized, Masked, Controlled, Safety and Efficacy Study of a Fluocinolone Acetonide Intravitreal Insert in Subjects With Chronic Non-Infectious Uveitis Affecting the Posterior Segment of the Eye
Brief Title: Safety and Efficacy of an Injectable Fluocinolone Acetonide Intravitreal Insert
Acronym: FAI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PSV-FAI-001
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Non-Infectious Uveitis
MeSH Terms: interventions — Bulk Drugs; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- sham injection (Sham Comparator): sham injection
  Interventions: Drug: Sham injection
- FAI insert (Experimental): FAI insert (0.18 mg fluocinolone acetonide)
  Interventions: Drug: FAI insert

INTERVENTIONS:
Drug: FAI insert
  Other Names: Active Drug
  Arms: FAI insert
Drug: Sham injection
  Other Names: Sham Comparator
  Arms: sham injection

SUMMARY:
A study to evaluate the safety and efficacy of an FAI insert for the management of subjects with non-infectious uveitis affecting the posterior segment of the eye.

DETAILED DESCRIPTION:
This is a phase 3, multi-national, multi-center, randomized, masked, controlled study to evaluate the safety and efficacy of an injectable fluocinolone acetonide intravitreal (FAI) insert for the management of subjects with non-infectious uveitis affecting the posterior segment of the eye. Patients will be randomized to receive either a sham injection or the FAI insert and will be observed for three years following treatment.

ELIGIBILITY:
Inclusion Criteria

* Male or non-pregnant female at least 18 years of age at time of consent
* One or both eyes having a history of recurrent non-infectious uveitis affecting the posterior segment of the eye with or without anterior uveitis > 1 year duration.
* During the 12 months prior to enrollment (Day 1), the study eye has either received treatment:
* systemic corticosteroid or other systemic therapies given for at least 3 months, and/or
* at least 2 intra- or peri-ocular injections of corticosteroid for management of uveitis

OR the study eye has experienced recurrence:

* at least 2 separate recurrences of uveitis requiring systemic, intra- or peri-ocular injection of corticosteroid
* At the time of enrollment (Day 1), study eye has < 10 anterior chamber cells/HPF and a vitreous haze ≤ grade 2.
* Visual acuity of study eye is at least 15 letters on the ETDRS chart
* Subject is not planning to undergo elective ocular surgery during the study
* Subject has ability to understand and sign the Informed Consent Form
* Subject is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria

* Allergy to fluocinolone acetonide or any component of the FAI insert
* History of posterior uveitis only that is not accompanied by vitritis or macular edema
* History of iritis only and no vitreous cells, anterior chamber cells or vitreous haze
* Uveitis with infectious etiology
* Vitreous hemorrhage
* Intraocular inflammation associated with a condition other than noninfectious uveitis (e.g. intraocular lymphoma)
* Ocular malignancy in either eye, including choroidal melanoma
* Toxoplasmosis scar in study eye; or scar related to previous viral retinitis
* Previous viral retinitis
* Current viral diseases of the cornea and conjunctiva including epithelial herpes simplex keratitis (dendritic keratitis), vaccinia, and varicella, mycobacterial infections of the eye or fungal diseases of ocular structure
* Media opacity precluding evaluation of retina and vitreous
* Peripheral retinal detachment in area of insertion
* Diagnosis of any form of glaucoma or ocular hypertension in study eye at Screening, unless study eye has been previously treated with an incisional surgery procedure that has resulted in stable IOP in the normal range (10-21 mmHg)
* Intraocular pressure (IOP) > 21 mmHg or concurrent therapy at screening with any IOP-lowering pharmacologic agent in the study eye
* Chronic hypotony (< 6 mmHg)
* Ocular surgery on the study eye within 3 months prior to study Day 1
* Capsulotomy in study eye within 30 days prior to study Day 1
* Prior intravitreal treatment of study eye with Retisert within 36 months prior to study Day 1
* Prior intravitreal treatment of study eye with Ozurdex within 6 months prior to study Day 1
* Prior intravitreal treatment of study eye with Triesence or Trivaris within 3 months prior to study Day 1
* Prior peri-ocular or subtenon steroid treatment of study eye within 3 months prior to study Day 1
* Subjects requiring chronic systemic or inhaled corticosteroid therapy (>15mg prednisone daily) or chronic systemic immunosuppressive therapy
* Excluding certain skin cancers (specifically, basal cell carcinoma and squamous cell carcinoma), any malignancy receiving treatment, or in remission less than 5 years prior to study Day 1
* Subjects who test positive for human immune deficiency virus (HIV) or syphilis during screening
* Mycobacterial uveitis or chorio-retinal changes of either eye which, in the opinion of the Investigator, result from infectious mycobacterial uveitis
* Systemic infection within 30 days prior to study Day 1
* Any severe acute or chronic medical or psychiatric condition that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, could make the subject inappropriate for entry into this study
* Any other systemic or ocular condition which, in the judgment of the investigator, could make the subject inappropriate for entry into this study
* Treatment with an investigational drug or device within 30 days prior to study Day 1
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from at least 14 days prior to study Day 1 until the Month 12 Visit
* Subjects unlikely to comply with the study protocol or who are likely to be lost to follow-up within three years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Jaffe, MD, Principal Investigator — Duke University Eye Center
Locations (34):
- United States (16):
  - Retina Vitreaous Associates, Beverly Hills, California
  - Retinal Consultants Medical Group, Inc, Sacramento, California
  - Retina Macula Institute, Torrance, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Northwestern University, Chicago, Illinois
  - Ophthalmology & Visual Sciences, Lexington, Kentucky
  - Ocular Immunology and Uveitis Foundation, Cambridge, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Retina Consultants, Slingerlands, New York
  - Duke University Eye Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OHSU Casey Eye Institute, Portland, Oregon
  - Charleston Neuroscience Institute, Ladson, South Carolina
  - Texas Retina Associates, Arlington, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Foresight Studies, LLC, San Antonio, Texas
- Germany (2):
  - Augenarzte am St. Franziskus Hospital, Münster
  - Universitatsklinikum Tubingen, Tübingen
- Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest, Hungary
- India (6):
  - L. V. Prasad Eye Institute - Hospital, Hyderabad, Andhra Pradesh
  - L.V. Prasad Eye Institute, Pātia, Bhubaneshwar
  - C.H Nagri Municipal Eye Hospital, Ahmedabad, Gujarat
  - Seth G.S. Medical College & KEM Hospital, Pārel, Mumbai
  - PBMA'S H.V. Desai Eye Hospital, Hadapsar, Pune
  - King George's Medical University, Lucknow, Uttar Pradesh
- Israel (3):
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Qiryat Ono
- United Kingdom (6):
  - Royal Hospitals Trust, Belfast
  - Birmingham and Midland Eye Centre, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Gloucestershire Royal Hospital, Gloucester
  - Moorfields Eye Hospital, London
  - St Thomas Hospital, London

REFERENCES:
- [Derived] Jaffe GJ, Pavesio CE; Study Investigators. Effect of a Fluocinolone Acetonide Insert on Recurrence Rates in Noninfectious Intermediate, Posterior, or Panuveitis: Three-Year Results. Ophthalmology. 2020 Oct;127(10):1395-1404. doi: 10.1016/j.ophtha.2020.04.001. Epub 2020 Apr 17. PMID 32624244

RESULTS

PARTICIPANT FLOW:
Groups:
- FAI Insert: FAI insert (0.18 mg fluocinolone acetonide)
  FAI insert
Period: Overall Study
Arm/Group | Sham Injection | FAI Insert
Started | 42 (Two investigators each site Investigator 1 unmasked treating and investigator 2 masked follow up.) | 87 (Two investigators each site Investigator 1 unmasked treating and investigator 2 masked follow up.)
Completed | 36 (Two investigators each site Investigator 1 unmasked treating and investigator 2 masked follow up.) | 80 (Two investigators each site Investigator 1 unmasked treating and investigator 2 masked follow up.)
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Population: A total of 129 (100%) subjects were included in the ITT and safety populations. 87 subjects in the FAI Insert 42 subjects in the Sham Injection
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Injection | FAI Insert | Total
Number analyzed (Participants) | 42 | 87 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (13.71) | 48.3 (13.90) | 48.3 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 50 | 79
  Male | 13 | 37 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 21 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 26 | 60 | 86
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hungary | 1 | 0 | 1
  United States | 19 | 37 | 56
  United Kingdom | 4 | 16 | 20
  Israel | 4 | 6 | 10
  Germany | 3 | 8 | 11
  India | 11 | 20 | 31
ITT and Safety populations [Count of Participants; unit: Participants]
  ITT | 42 | 87 | 129
  Safety | 42 | 87 | 129

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Recurrence of Uveitis in the Study Eye and Overall Summary of Number of Participants With Ocular Treatment-Emergent Adverse Events for the Study Eye Through Month 36 Visit
Description: Safety: Ocular adverse events, including IOP elevation; medications/procedures required to control elevated IOP; development or worsening of cataract; cataract-related procedures; clinically significant ocular changes; procedure related adverse events Primary Efficacy Endpoint: Proportion of subjects who have a recurrence of uveitis in the study eye within 6 months after receiving study treatment.
Time Frame: 36 months
Population: Proportion of Subjects with Recurrence of Uveitis in the Study Eye at 36 Months (ITT Population)
  Overall Summary of Ocular Treatment-Emergent Adverse Events for the Study Eye Through Month 36 Visit (Safety Population)
Measure: Count of Participants; unit: Participants
Groups:
- Sham Injection: sham injection
  Sham injection The sham applicator was an empty 1-mL syringe attached to a blunt 14-gauge needle; it did not contain an FAI insert. During study Day 1, the sham applicator was gently pressed against the study eye to provide the subject with the perception that an intravitreal injection was being performed. This procedure was performed to mask study subjects to their assigned treatment.
- FAI Insert: FAI insert (0.18 mg fluocinolone acetonide) One treatment (FAI injection) was administered on Day 1 to each subject. The Fluocinolone Acetonide Intravitreal Insert (FAI insert) is an injectable intravitreal sustained-release FA delivery system preloaded into an injection device. Each insert contained a drug core of FA as the active ingredient within a cylindrical polyimide polymer tube 3.5-mm long with an external diameter of 0.37 mm.
  The dose delivered in the FAI insert was 0.18 mg fluocinolone acetonide delivered into the vitreous humor for 36 months. The FAI insert was administered to the study eye by injection through the pars plana using a preloaded applicator with a 25-gauge needle.
Arm/Group | Sham Injection | FAI Insert
Number analyzed (Participants) | 42 | 87
Participants
  Protocol-Defined Recurrence of Uveitis | 12 | 5
  Ocular TEAE | 39 | 77
  Ocular Serious TEAE | 12 | 16
  Ocular Treatment- Related TEAE | 21 | 60
  Ocular Treatment-Related Serious TEAE | 2 | 11
  Ocular TEAE leading to treatment discontinuation | 0 | 0
  Ocular TEAE leading to study discontinuation | 0 | 0
  Ocular AE leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Treatment-Emergent Non-Ocular Adverse Events Through Month 36 Visit by System Organ Class and Preferred Term, Greater than 5% of Subjects in Either Treatment Group (Safety Population)
Arm/Group | Sham Injection | FAI Insert
All-Cause Mortality (participants affected / at risk) | 0/42 | 1/87
Serious Adverse Events (participants affected / at risk) | 17/42 | 29/87
Other Adverse Events (participants affected / at risk) | 40/42 | 84/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sham Injection (N=42) | FAI Insert (N=87)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 7
Cystoid macular oedema (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 1
Hypotony of eye (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 2 | 0
Non-infectious endophthalmitis (Eye disorders) | 2 | 0
Ocular hypertension (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 4 | 2
Vitreous haemorrhage (Eye disorders) | 1 | 0
Vitritis (Eye disorders) | 0 | 1
Intraocular pressure fluctuation (Investigations) | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 2
Post-procedural inflammation (Injury, poisoning and procedural complications) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Injection (N=42) | FAI Insert (N=87)
Hypertension (Vascular disorders) | 4 (4) | 6 (6)
Intraocular pressure increased (Investigations) | 13 (13) | 28 (28)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 6 (6)
Anterior chamber flare (Eye disorders) | 3 (3) | 0 (0)
Cataract (Eye disorders) | 6 (6) | 33 (33)
Cataract subcapsular (Eye disorders) | 4 (4) | 6 (6)
Conjunctival haemorrhage (Eye disorders) | 5 (5) | 13 (13)
Cystoid macular oedema (Eye disorders) | 12 (12) | 12 (12)
Dry eye (Eye disorders) | 5 (5) | 15 (15)
Eye pain (Eye disorders) | 9 (9) | 11 (11)
Eye pruritus (Eye disorders) | 3 (3) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 5 (5)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 8 (8)
Iridocyclitis (Eye disorders) | 6 (6) | 1 (1)
Macular fibrosis (Eye disorders) | 5 (5) | 5 (5)
Macular oedema (Eye disorders) | 16 (16) | 6 (6)
Ocular discomfort (Eye disorders) | 1 (1) | 5 (5)
Ocular hyperaemia (Eye disorders) | 5 (5) | 7 (7)
Photopsia (Eye disorders) | 3 (3) | 5 (5)
Posterior capsule opacification (Eye disorders) | 3 (3) | 5 (5)
Uveitis (Eye disorders) | 26 (26) | 18 (18)
Vision blurred (Eye disorders) | 3 (3) | 2 (2)
Visual acuity reduced (Eye disorders) | 5 (5) | 16 (16)
Visual impairment (Eye disorders) | 3 (3) | 8 (8)
Vitreous floaters (Eye disorders) | 5 (5) | 8 (8)
Vitreous opacities (Eye disorders) | 4 (4) | 2 (2)
Fatigue (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 3 (3) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3)
Hypothyroidism (Endocrine disorders) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 12 (12)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Conjunctivitis (Infections and infestations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT01694186/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/86/NCT01694186/SAP_001.pdf